CLINICAL TRIAL: NCT05181072
Title: Assessing the Effectiveness of Virtual Versus In-person Peer-motivation Smoking Cessation Interventions
Brief Title: Identify the Usefulness of In-person and Virtual Quit Smoking Programs
Acronym: CEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morgan State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Payam Sheikhattari, Professor, Morgan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: #19/06-0082; 5U54MD013376 (NIH)
Record Dates: First submitted 2021-08-19; First posted 2022-01-06 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Cigarette Smoking; Tobacco Use
Keywords: Smoking cessation program; Community-based participatory research; Peer-based approach; underserved population
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced in-person peer-motivation (Experimental): This is a seven-week tobacco cessation program and will be offered in-person weekly for seven weeks and will utilize the CEASE Today Tobacco Cessation Manual.
  Interventions: Behavioral: Enhanced in-person peer-motivation smoking cessation
- Virtual peer-motivation (Experimental): This is a seven-week tobacco cessation program and will be offered virtually (except first two sessions: orientation and technology set-up) weekly for seven weeks and will utilize a newly developed website with smoking cessation modules that mirrors lessons of the CEASE Today Tobacco Cessation Manual.
  Interventions: Behavioral: Virtual peer-motivation smoking cessation
- Self-help/Control (No Intervention): The participants in the control group will receive the services already in place, including a brief motivation enhancement session.

INTERVENTIONS:
Behavioral: Enhanced in-person peer-motivation smoking cessation — Tobacco cessation classes will be offered in-person for a total of five sessions delivered weekly for five weeks and will utilize the CEASE Today Tobacco This is a seven-week tobacco cessation program and will be offered in-person weekly for seven weeks and will utilize the CEASE Today Tobacco Cessation Manual.
  Arms: Enhanced in-person peer-motivation
Behavioral: Virtual peer-motivation smoking cessation — This is a seven-week tobacco cessation program and will be offered virtually (except first two sessions: orientation and technology set-up) weekly for seven weeks and will utilize a newly developed website with smoking cessation modules that mirrors lessons of the CEASE Today Tobacco Cessation Manual
  Arms: Virtual peer-motivation

SUMMARY:
This study is a randomized community-based trial adapted to the needs of adults aged 21 years or older that is designed by an existing research partnership called Communities Engaged and Advocating for Smoke-free Environments (CEASE). The overarching goal of the proposed study is to apply a community-based approach to reduce tobacco use among low-income communities in Baltimore City. The study setting represents three underserved communities in Baltimore City: the Oldtown/Middle East, the Waverlies, Poppleton/The Terraces/Hollins Market, and Washington Village/Pigtown. Poppleton/The Terraces/Hollins Market and Washington Village/Pigtown will be considered as one community. The three communities have been randomly allocated to one of the three arms of the study: 1) Virtual intervention, 2) Enhanced in-person intervention, and 3) The control community.

The Waverlies was assigned to virtual, the Middle East was assigned to be the in-person group, and Poppleton/The Terraces/Hollins Market and Washington Village/Pigtown became the self-help/control group. The goal of the trial is to assess the effectiveness of virtual versus in-person versions of a smoking cessation program in terms of their success rates (quitting and staying quit). The study's primary hypothesis is that the smoking cessation rate will be equal to or higher in the virtual peer-motivation arm than the in-person and self-help/ control arms. The secondary hypothesis is that the retention rate will differ among the three interventions (virtual peer-motivation, enhanced in-person peer-motivation, and self-help/control community).

Virtual and enhanced in-person versions of the CEASE Today Peer-Motivation Intervention were developed and pilot-tested during the first and second years based on local data and input from partnering communities. The enhanced in-person intervention will utilize the existing CEASE Today Tobacco Cessation Manual with improvements. The virtual intervention will use a newly developed CEASE website with smoking cessation modules and lessons that mirror the CEASE Today Tobacco Cessation Manual. Trained peer-motivators will deliver the intervention and be actively involved in recruiting the participants, motivation enhancement, group facilitation, and counseling.

DETAILED DESCRIPTION:
The project will capitalize on the capacity of a long-term successful community-campus partnership to reduce tobacco-related health disparities through a mixed-method randomized community-based trial adapted to the needs of adults (>21 y/o). The smoking cessation classes will be conducted in community venues, including non-profit organizations, churches, schools, etc., in three underserved communities in Baltimore City. The three communities have been randomly allocated to one of the three arms of the study:

1. Enhanced in-person intervention
2. Virtual intervention
3. The self-help/control community

CEASE Digital smoking cessation program is a seven-week program using the CEASE Today Tobacco cessation manual. Sessions during the first two weeks will be held in-person for both the virtual and enhanced in-person arms after which the subsequent sessions will be conducted either virtually or in-person for the respective arms. Week one will entail an orientation session. Following the screening, all eligible participants will be invited to the orientation session where the participants will be taken through the informed consent process. After completing the informed consent process, each participant will complete a baseline survey and take a carbon monoxide (CO) breath test. The participants will be given relevant introductory information about the CEASE Digital program.

In addition, participants will be given one month/30 days to set a quit date and will receive Nicotine Replacement Therapy (NRT) samples along with information about using NRT. Orientation packets, with relevant materials, will be provided to the participants and intervention site coordinators. In the second week, which will also be held in-person for all the participants, class information and technology training (using zoom and slack) will be provided. Participants will get an opportunity to practice accessing the program materials and /curriculum via the digital platforms. In addition, ground rules for the meetings will be set, including group meeting etiquette and maintaining confidentiality.

CEASE Today Tobacco Cessation program will commence in week three and will continue for a total of five sessions delivered weekly for five weeks. Smoking cessation classes (support groups) will be delivered either in-person or virtually. Each session will last for 2 hours, and trained peer-motivators will deliver the classes. Participants will be enrolled in groups of up to 10-15 individuals.

The enhanced in-person intervention will utilize the CEASE Today Tobacco Cessation Manual. Different topics from the manual will be covered in each session, and participants will engage in discussion regarding the respective topics. Several activities will be conducted related to the session topics during each session to ensure the active participation of the program participants and the understanding and retention of the information provided. In addition, the participants will be given assignments at the end of each session to keep them engaged and motivated in between classes.

For the virtual intervention, a newly developed website with smoking cessation modules will be used that mirror lessons of the CEASE Today Tobacco Cessation Manual. In this arm, participants are given access to the CEASE website and provided with virtual materials, information, and resources by their assigned peer motivators. Virtual smoking cessation peer motivation sessions are offered using the digital online platform zoom. Participants in the virtual group form closed groups and will communicate with their group mates and peer-motivators through email and text messages throughout the intervention. Different topics will be covered in each session, and participants will engage in discussion regarding the respective topics (please see appendix 13 for more details). In addition, the participants will be given assignments at the end of each session to keep them engaged and motivated in between classes.

From week three during each session, the participants will be given the weekly check-in form to complete. All participants will be followed approximately three months after their completion of smoking cessation classes to ascertain their smoking status and will complete the follow-up survey and CO breath test.

The participants in the self-help/control group will receive the services already in place, including a brief motivation enhancement session. They will also receive a brief peer motivation and orientation to self-help smoking cessation materials (hard copy of CEASE Today Tobacco Cessation Manual and the link to the CEASE web materials), other available resources including information about the local tobacco cessation services available. The participants in the self-help/control group will complete the follow-up survey and CO breath test three months after enrollment.

The sample calculation was performed based on the primary outcome variable (smoking cessation) using statistical software Stata. Based on the previous experience with the CEASE smoking cessation program, it can be assumed that the quit rates for the virtual, in-person, and self-help/control groups will be approximately in the ranges of 8-20%, 10-25%, and 3-12%, respectively. Therefore, the goal is to enroll 210 Adults in each of the three arms of the study with a total planned enrollment of 630 individuals over two years. This will give enough power to document a difference in smoking cessation/ abstinence rate of (5% - 8%) between groups.

The data will be exported from KoBoToolbox as an excel file and will be imported to statistical software Stata for cleaning and analysis. The descriptive univariate analysis will be done to review each variable and summarize demographic information. The result will be presented as mean and standard deviation for continuous variables and percentage for categorical variables. The bivariate analysis will be done to compare quit rates with some potential predictor variables using Chi-square tests of independence for categorical variables (gender, race, education, employment) and Student's T-test for continuous variables (age and Fagerstrom score). The results will be presented as numbers with corresponding proportions for the Chi-square tests and presented as means with standard deviations for the T-tests.

To handle missing data at follow-up, analysis of the primary outcome will be done in two scenarios. In one scenario, participants with missing outcome data will be considered as still smoking and will therefore be included in the analysis. This will give the worst case scenario of quit rates in the study population. In the second scenario, only participants who responded to the survey will be included in the analysis. For other variables with missing data, records will be deleted if missing data is over 90% and if less than 90%, the missing data will be left out of the analysis of each variable.

Data will be primarily collected by trained peer-motivators at the intervention sites under the supervision of the research staff. The principal investigator and the research scientist provide technical and logistical support to peer motivators and assume the overall responsibility for the accuracy, completeness, legibility, and timeliness of the collected data. All source documents will be completed in a neat, legible manner to ensure accurate interpretation of data.

Hardcopies of the study visit worksheets will be provided for use as source document worksheets for recording data for each participant enrolled in the study. Data recorded in the electronic form derived from source documents should be consistent with the data recorded on the source documents. The collected data will be exported from KoBoToolbox as an excel file and will be imported to statistical software Stata for cleaning and analysis and in compliance with 21 CFR Part 11-compliant data capture system. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Clinical data will be entered directly from the source documents.

Each intervention site will be overseen for quality assurance and quality control purposes to maintain the integrity of research, data collection, documentation, and completion activities. Quality control (QC) measures will be implemented beginning with the data entry system followed by checking the accuracy of collected data and preparing the database for analyses. Any missing data or data anomalies will be checked by the research scientist and communicated to the site(s) and/or the peer motivator(s) for clarification/resolution. The research scientist will follow and review the Standard Operating Procedures (SOPs) and CEASE Digital Data Management and Quality Assurance documents developed to evaluate and verify that the clinical trial is conducted and data are collected, documented (recorded), and reported in compliance with the protocol, ethical standards, regulatory compliance, and accuracy. The study's senior research associate will review the informed consent forms, survey questionnaires, weekly check-in forms, and follow-up survey questionnaires for accuracy.

The research staff will be provided direct access to relevant source data/documents, and reports for the purpose of monitoring, auditing, and inspecting potential data irregularities and/or inaccuracies. The PI and the senior research associate oversee the overall research, data collection, and documentation activities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 21 years and above
* Current smokers
* Willing and ready to quit using tobacco, and consent to participate
* Access to devices (desktop, laptop, tablets, etc) with reliable and consistent internet access or cellular data (to participate in the virtual intervention)

Exclusion Criteria:

* Individuals who have health conditions preventing them from providing consent
* Individuals in communities randomized to the virtual intervention with no access to smartphones with internet access or cellular data

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Self-reported smoking cessation verified by expired-air Carbon Monoxide (CO) level (virtual and in-person groups). | week19 from enrollment (12 weeks after the last peer-motivation session)
  Self-reported smoking cessation verified by expired-air Carbon Monoxide (CO) levels. This will be measured using the CO breath monitor. Levels less than 8ppm will be considered as quit.
Self-reported smoking cessation verified by expired-air Carbon Monoxide (CO) level (self-help group). | week12 from enrollment
  Self-reported smoking cessation verified by expired-air Carbon Monoxide (CO) levels. This will be measured using the CO breath monitor. Levels less than 8ppm will be considered as quit.

SECONDARY OUTCOMES:
Retention | Week 7
  Retention will be measured by the number of in-person or virtual sessions attended

CONTACTS AND LOCATIONS:
Locations (1):
- Morgan CARES, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burns EK, Deaton EA, Levinson AH. Rates and reasons: disparities in low intentions to use a state smoking cessation quitline. Am J Health Promot. 2011 May-Jun;25(5 Suppl):S59-65. doi: 10.4278/ajhp.100611-QUAN-183. PMID 21510788
- [Background] Cummings KM, Orleans CT. Policies to Achieve a Smoke-Free Society: A Research Agenda for 2010-2015. 2009.
- [Background] Cavazos-Rehg PA, Breslau N, Hatsukami D, Krauss MJ, Spitznagel EL, Grucza RA, Salyer P, Hartz SM, Bierut LJ. Smoking cessation is associated with lower rates of mood/anxiety and alcohol use disorders. Psychol Med. 2014 Sep;44(12):2523-35. doi: 10.1017/S0033291713003206. PMID 25055171
- [Background] Henry SA., Sheikhattari P, Wagner FA. Analyzing disparities on tobacco use through CBPR. Drug & Alcohol Dependence. 2015; 146, p. e140.
- [Background] Ford P, Clifford A, Gussy K, Gartner C. A systematic review of peer-support programs for smoking cessation in disadvantaged groups. Int J Environ Res Public Health. 2013 Oct 28;10(11):5507-22. doi: 10.3390/ijerph10115507. PMID 24169412
- [Background] McKay CE, Dickerson F. Peer Supports for Tobacco Cessation for Adults with Serious Mental Illness: A Review of the Literature. J Dual Diagn. 2012;8(2):104-112. doi: 10.1080/15504263.2012.670847. Epub 2012 May 11. PMID 22904697
- [Background] O'Toole TP, Aaron KF, Chin MH, Horowitz C, Tyson F. Community-based participatory research: opportunities, challenges, and the need for a common language. J Gen Intern Med. 2003 Jul;18(7):592-4. doi: 10.1046/j.1525-1497.2003.30416.x. No abstract available. PMID 12848844
- [Background] Wallerstein N, Duran B, Oetzel JG, Minkler M. Community-Based Participatory Research for Health: Advancing Social and Health Equity, John Wiley & Sons. 2017.
- [Background] Prado GF, Lombardi EM, Bussacos MA, Arrabal-Fernandes FL, Terra-Filho M, Santos Ude P. A real-life study of the effectiveness of different pharmacological approaches to the treatment of smoking cessation: re-discussing the predictors of success. Clinics (Sao Paulo). 2011;66(1):65-71. doi: 10.1590/s1807-59322011000100012. PMID 21437438
- [Background] Jain A. Treating nicotine addiction. BMJ. 2003 Dec 13;327(7428):1394-5. doi: 10.1136/bmj.327.7428.1394. No abstract available. PMID 14670889
- [Background] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. The Health Consequences of Smoking-50 Years of Progress: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK179276/ PMID 24455788
- [Background] Raw M, McNeill A, West R. Smoking cessation: evidence based recommendations for the healthcare system. BMJ. 1999 Jan 16;318(7177):182-5. doi: 10.1136/bmj.318.7177.182. No abstract available. PMID 9888919
- [Background] Ramo DE, Liu H, Prochaska JJ. A mixed-methods study of young adults' receptivity to using Facebook for smoking cessation: if you build it, will they come? Am J Health Promot. 2015 Mar-Apr;29(4):e126-35. doi: 10.4278/ajhp.130326-QUAL-128. Epub 2014 Feb 27. PMID 24575728
- [Background] Ranney L, Melvin C, Lux L, McClain E, Lohr KN. Systematic review: smoking cessation intervention strategies for adults and adults in special populations. Ann Intern Med. 2006 Dec 5;145(11):845-56. doi: 10.7326/0003-4819-145-11-200612050-00142. Epub 2006 Sep 5. PMID 16954352
- [Background] Elfeddali I, Bolman C, Candel MJ, Wiers RW, De Vries H. The role of self-efficacy, recovery self-efficacy, and preparatory planning in predicting short-term smoking relapse. Br J Health Psychol. 2012 Feb;17(1):185-201. doi: 10.1111/j.2044-8287.2011.02032.x. Epub 2011 Jun 27. PMID 22107073
- [Background] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Background] Cokkinides VE, Ward E, Jemal A, Thun MJ. Under-use of smoking-cessation treatments: results from the National Health Interview Survey, 2000. Am J Prev Med. 2005 Jan;28(1):119-22. doi: 10.1016/j.amepre.2004.09.007. PMID 15626567
- [Background] Cokkinides VE, Halpern MT, Barbeau EM, Ward E, Thun MJ. Racial and ethnic disparities in smoking-cessation interventions: analysis of the 2005 National Health Interview Survey. Am J Prev Med. 2008 May;34(5):404-12. doi: 10.1016/j.amepre.2008.02.003. PMID 18407007
- [Background] West R, Sohal T. "Catastrophic" pathways to smoking cessation: findings from national survey. BMJ. 2006 Feb 25;332(7539):458-60. doi: 10.1136/bmj.38723.573866.AE. Epub 2006 Jan 27. PMID 16443610
- [Background] Orleans CT. Increasing the demand for and use of effective smoking-cessation treatments reaping the full health benefits of tobacco-control science and policy gains--in our lifetime. Am J Prev Med. 2007 Dec;33(6 Suppl):S340-8. doi: 10.1016/j.amepre.2007.09.003. PMID 18021909
- [Background] Blanco C, Olfson M, Goodwin RD, Ogburn E, Liebowitz MR, Nunes EV, Hasin DS. Generalizability of clinical trial results for major depression to community samples: results from the National Epidemiologic Survey on Alcohol and Related Conditions. J Clin Psychiatry. 2008 Aug;69(8):1276-80. doi: 10.4088/jcp.v69n0810. PMID 18557666
- [Background] Peek ST, Wouters EJ, van Hoof J, Luijkx KG, Boeije HR, Vrijhoef HJ. Factors influencing acceptance of technology for aging in place: a systematic review. Int J Med Inform. 2014 Apr;83(4):235-48. doi: 10.1016/j.ijmedinf.2014.01.004. Epub 2014 Jan 19. PMID 24529817
- [Background] Gücin NÖ, Berk ÖS. Technology Acceptance in Health Care: An Integrative Review of Predictive Factors and Intervention Programs. 2015. Procedia - Social and Behavioral Sciences, 195, pp. 1698-1704.
- [Background] Wang TW, Gentzke A, Sharapova S, Cullen KA, Ambrose BK, Jamal A. Tobacco Product Use Among Middle and High School Students - United States, 2011-2017. MMWR Morb Mortal Wkly Rep. 2018 Jun 8;67(22):629-633. doi: 10.15585/mmwr.mm6722a3. PMID 29879097
- [Background] Centers for Disease Control and Prevention (CDC). Tobacco product use among middle and high school students--United States, 2011 and 2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 15;62(45):893-7. PMID 24226625
- [Background] Corey CG, Ambrose BK, Apelberg BJ, King BA. Flavored Tobacco Product Use Among Middle and High School Students--United States, 2014. MMWR Morb Mortal Wkly Rep. 2015 Oct 2;64(38):1066-70. doi: 10.15585/mmwr.mm6438a2. PMID 26421418
- [Background] Wagner FA, Sheikhattari P, Buccheri J, Gunning M, Bleich L, Schutzman C. A Community-Based Participatory Research on Smoking Cessation Intervention for Urban Communities. J Health Care Poor Underserved. 2016;27(1):35-50. doi: 10.1353/hpu.2016.0017. PMID 27763459
- [Background] Sheikhattari P, Zhu S, Clubb P, Wagner FA. New insights on tobacco smoking among underserved and poor. 2010: pp. 400-405.
- [Background] Sheikhattari P, Apata J, Kamangar F, Schutzman C, O'Keefe A, Buccheri J, Wagner FA. Examining Smoking Cessation in a Community-Based Versus Clinic-Based Intervention Using Community-Based Participatory Research. J Community Health. 2016 Dec;41(6):1146-1152. doi: 10.1007/s10900-016-0264-9. PMID 27688221
- [Background] Estreet A, Apata J, Kamangar F, Schutzman C, Buccheri J, O'Keefe AM, Wagner F, Sheikhattari P. Improving Participants' Retention in a Smoking Cessation Intervention Using a Community-based Participatory Research Approach. Int J Prev Med. 2017 Dec 19;8:106. doi: 10.4103/ijpvm.IJPVM_303_17. eCollection 2017. PMID 29416835
- [Background] Cheung KL, de Ruijter D, Hiligsmann M, Elfeddali I, Hoving C, Evers SMAA, de Vries H. Exploring consensus on how to measure smoking cessation. A Delphi study. BMC Public Health. 2017 Nov 21;17(1):890. doi: 10.1186/s12889-017-4902-7. PMID 29162043
- [Background] Moberg J, Kramer M. A brief history of the cluster randomised trial design. J R Soc Med. 2015 May;108(5):192-8. doi: 10.1177/0141076815582303. No abstract available. PMID 26022551
- [Background] Wagner F, Sheikhattari P. 1968 - Improving the retention rates of two evidence-based smoking cessation trials designed through a participatory approach. European Psychiatry. 2013; 28(Supplement 1), p. 1.
- [Background] Fagerstrom KO, Schneider NG. Measuring nicotine dependence: a review of the Fagerstrom Tolerance Questionnaire. J Behav Med. 1989 Apr;12(2):159-82. doi: 10.1007/BF00846549. PMID 2668531
- [Background] Broadhead WE, Gehlbach SH, de Gruy FV, Kaplan BH. The Duke-UNC Functional Social Support Questionnaire. Measurement of social support in family medicine patients. Med Care. 1988 Jul;26(7):709-23. doi: 10.1097/00005650-198807000-00006. PMID 3393031
- See also: Burden of Tobacco Use in the U.S. — https://www.cdc.gov/tobacco/campaign/tips/resources/data/cigarette-smoking-in-united-states.html